CLINICAL TRIAL: NCT03543384
Title: Imaging of Facial Neuritis Using T2-weighted Gradient-echo Fast Imaging Employing Steady State Acquisition After Gadolinium Injection
Brief Title: Imaging of Facial Neuritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6810
Record Dates: First submitted 2018-02-26; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-02

CONDITIONS: Facial Neuritis
Keywords: facial neuritis; T2 weighted gradient-echo; fast imaging employing steady state acquisition (FIESTA-C); magnetic resonance imaging (MRI)
MeSH Terms: conditions — Facial Nerve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Improved means of positive diagnosis of facial neuritis, the leading cause of peripheral facial palsy

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Subject giving their consent for their participation
* Patients with neuritis facial (neuritis group) who benefited, between 2009 and 2016, from an MRI of the internal auditory ducts, with gadolinous product injection and on the MRI 3 Tesla
* Patients with a perception deafness, without neuritis sign (control group) who also benefited from an MRI with gadolinous product injection on the MRI 3T with the same protocol.

Exclusion Criteria:

- Refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with neuritis facial (neuritis group) who benefited, between 2009 and 2016, from an MRI of the internal auditory ducts, with gadolinous product injection and on the MRI 3 Tesla
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of pathologic enhancement of the facial nerve on the symptomatological side of the T2 sequence (FIESTA-C) | 1 hour after the realization of the MRI

CONTACTS AND LOCATIONS:
Overall Officials: Francis VEILLON, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service Imagerie 1, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No